CLINICAL TRIAL: NCT05662306
Title: Comprehensive Treatment of Early Course Schizophrenia: A Nonrandomized Study of Long Acting Injectable Antipsychotic Medication Combined With Cognitive and Functional Skills Training
Brief Title: C-Cog in Early Course Schizophrenia Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: University of Miami (Other)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Principal Investigator, Dante Durand, Associate Professor of Psychiatry, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20211098
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
Keywords: Relapse; Remission; Recovery
MeSH Terms: conditions — Schizophrenia; Recurrence | interventions — aripiprazole lauroxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aripiprazole and Computerized Cognitive and Functional Skills Training Group (Experimental): Participants in this arm will receive long-acting injectable aripiprazole every 2 months formulation for 12 consecutive months. Participants in this arm will also receive Computerized cognitive and functional skills training during the first 12 weeks of study participation.
  Interventions: Drug: Aripiprazole Lauroxil; Behavioral: Computerized cognitive and functional skills training

INTERVENTIONS:
Drug: Aripiprazole Lauroxil — 1064 mg 2-month long-acting injectable administered as an intramuscular injection over a 12-month period.
Behavioral: Computerized cognitive and functional skills training — Self-administered cognitive and technology focused skills training, administered at home for 2 hours per week for the first 12 weeks of the 12-month study period.

SUMMARY:
The purpose of this study is to examine the role of clinical stability in functional recovery. in first episode schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Adults
2. Diagnosis of schizophrenia
3. Current Hospitalization or outpatient relapse
4. Fewer than four previous admissions
5. Willing to accept long-acting injectable treatment and participate in rehabilitation

Exclusion Criteria:

1. Primary diagnosis other than schizophrenia
2. Prior Long Acting Injectable treatment
3. Current Suicide Risk
4. Hypersensitivity to Aripiprazole
5. Pregnancy
6. Positive illicit drug screen other than cannabis (rescreening allowed in 4 weeks for drug positive cases)
7. Unable to give personal informed consent
8. History of treatment resistance as evidenced by clozapine treatment
9. Unable to stop treatment with medications that are strong Cytochrome (CYP) 2D6 or CYP 3A4 inhibitors and or strong CYP3A4 inducers (2.3, 7.1) for at 14 days prior to initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dante Durand, MD, Principal Investigator — University of Miami Miller School
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aripiprazole and Computerized Cognitive and Functional Skills Training Group
Started | 1
Completed | 0
Not Completed | 1
Not completed — Sponsor terminated and PI withdrew participant | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aripiprazole and Computerized Cognitive and Functional Skills Training Group
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Who Develop Sustained Remission of Symptoms of Schizophrenia as Measured as Having a Score of 3 or Less on All 6 Critical Items From the Positive and Negative Syndrome Scale (PANSS)
Description: PANSS has 6 critical items with each item being scored from 1 to 7 with the higher score indicating more severe symptoms. A score of 3 or less on all six critical items defines the presence of remission.
Time Frame: 6 months
Measure: Number; unit: Percentage of participants
Arm/Group | Aripiprazole and Computerized Cognitive and Functional Skills Training Group
Number analyzed (Participants) | 1
Percentage of participants | 100

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Aripiprazole and Computerized Cognitive and Functional Skills Training Group
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT05662306/Prot_SAP_000.pdf